CLINICAL TRIAL: NCT02946190
Title: A Phase II Randomized, Observer-blind Controlled Pilot Study to Compare the Safety and Immunogenicity of Acellular Pertussis Vaccines Including Chemically or Genetically-detoxified Pertussis Toxin in Adolescents Aged 11-15 Years Previously Immunized With Acellular Pertussis Vaccines
Brief Title: The PertADO Geneva Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Siegrist Claire-Anne (Other)
Collaborators: BioNet-Asia Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Siegrist Claire-Anne, Director of Center for Vaccinology, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CER 2016-00500
Record Dates: First submitted 2016-10-24; First posted 2016-10-27 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Pertussis
Keywords: Acellular pertussis vaccines Genetically-detoxified pertussis toxin Adolescents
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Pertagen® aP + Td-pur® (Experimental): BioNet-Asia recombinant acellular Pertussis vaccine (Pertagen®) given simultaneously with Td-pur® vaccine (Novartis/GSK) intramuscularly as a single dose on Day 0
  Interventions: Biological: Pertagen® aP + Td-pur®
- Arm 2: Boostrix® dTpa (Active Comparator): Licensed Tetanus-diphtheria (reduced dose)-acellular Pertussis vaccine (Boostrix® dTpa; GSK) given intramuscularly as a single dose on Day 0
  Interventions: Biological: Boostrix® dTpa

INTERVENTIONS:
Biological: Pertagen® aP + Td-pur® — see arm/group descriptions
  Arms: Arm 1: Pertagen® aP + Td-pur®
Biological: Boostrix® dTpa — see arm/group descriptions
  Arms: Arm 2: Boostrix® dTpa

SUMMARY:
This is a phase II, randomized double-center, and observer-blind controlled pilot vaccine trial in 11 to 15 years old healthy subjects to assess the immunogenicity of the genetically detoxified pertussis toxin (rPT) included in a novel acellular pertussis vaccine (Pertagen®) manufactured by BioNet-Asia when delivered by the intramuscular route to adolescents previously primed and boosted with chemically-detoxified PT, along with Td-pur® and in comparison with that of Boostrix® dTpa.

At Day 0, eligible volunteers will undergo a venous bleed for the determination of baseline values and enter the randomization scheme, being allocated to one of two groups: A (Pertagen® + Td-pur®), B (Boostrix® dTpa).

Randomized participants will receive one dose of Pertagen® and Td-pur® (Group A) or 1 dose of Boostrix® dTpa (Group B) by intramuscular injection in the deltoid. All subjects will be observed in the Plateforme de Recherché Pédiatrique for 30 minutes after immunization.

Post-immunization local and systemic reactions will be followed up for 7 days after immunization. Adverse events will be followed for 28 days after immunization.

At Day 28, a second visit (study end visit) will take place for safety evaluation and blood draw for immunogenicity evaluation.

Blood draws performed on Day 0 (Baseline) and Day 28 will be used to evaluate immune response to study vaccines.

The primary statistical analysis will be performed with visit 2 (Day 28) data to compare the immunogenicity and safety of one dose of Pertagen®, given simultaneously with Td-pur®, to those elicited by Boostrix® dTpa.

DETAILED DESCRIPTION:
A significant increase of pertussis incidence is reported in a growing number of countries. This resurgence is considered as resulting from the limited durability of aP-vaccine-induced immunity and is associated with increased mortality in young infants and morbidity at all age groups. As the pertussis immunity acquired through immunization or infection is short-lived, its maintenance or reactivation requires repeat boosting at regular time points. Thus, novel strategies capable of reactivating pertussis immunity in older children, adolescents or adults, including pregnant women, are needed.

A puzzling observation is that the efficacy of current acellular pertussis vaccines (which contain chemically-detoxified pertussis toxoid (PT)) is higher in infants and children than adolescents, in whom vaccine efficacy is limited and rapidly wanes. This may derive - at least in part - from priming and repeat immunizations with acellular vaccines containing chemically-detoxified PT and thus induction of antibodies specific of the chemically-detoxified PT but unable to efficiently recognize the native PT expressed by B. pertussis.

The development of optimized acellular pertussis vaccines should thus include antigens with a similar immunogenicity profile as native PT but deprived of its toxic properties. This is best achieved through the genetic rather than chemical detoxification of PT, which results in both nontoxic and immunogenic PT.

Clinical studies have shown the good tolerability profile and the superior immunogenicity profile of acellular pertussis vaccines including genetically-detoxified PT (rPT) in adults and adolescents previously primed with whole-cell pertussis (wP) vaccines. As whole-cell vaccines express native PT, whether the superior immunogenicity of rPT will be observed in adolescents/adults previously primed with acellular pertussis vaccines containing chemically-detoxified PT is of key importance.

This is a phase II randomized, observer-blind controlled study to compare the safety and immunogenicity of acellular pertussis vaccines including chemically or genetically-detoxified pertussis toxin in adolescents aged 11-15 years. The primary objective is to assess the immunogenicity of the genetically detoxified pertussis toxin (rPT) included in a novel acellular pertussis vaccine (Pertagen®) when delivered by the intramuscular route to adolescents previously primed and boosted with chemically-detoxified PT, along with Td-pur® and in comparison with that of Boostrix® dTpa. The secondary objectives are (1) to assess safety of Pertagen® when administered with Td-pur® to adolescents as compared to Boostrix® dTpa and (2) to assess the humoral responses elicited by Pertagen® when administered with Td-pur® as compared to Boostrix® dTpa.

In this study, exploratory immunological measures will also be performed (pending sufficient or additional funding). These are anticipated to include:

* The assessment of antibody titers to specific neutralizing and non-neutralizing epitopes of PT, by competitive ELISA, before and after (Day 28) boosting with Pertagen® and Boostrix® dTpa.
* To assess cellular responses to PT before and after boosting with Pertagen® and Boostrix® dTpa.
* To assess the frequency and phenotype of PT-specific memory B cell responses (as compared to tetanus toxoid) before and after boosting with Pertagen® or Boostrix® dTpa (i.e. at Day 0 and Day 28).
* To characterize changes in cellular responses following boosting with Pertagen® or Boostrix® dTpa

Three vaccines will be used in the study. The BioNet-Asia study vaccine (Pertagen®), Td-pur® (Novartis/GSK) which will be concomitantly administered with the study vaccine, and the control Boostrix® dTpa.

The investigational product Pertagen® will be manufactured, labeled, packaged and released for clinical use by BioNet-Asia, in accordance with the requirements of Good Manufacturing Practices.Both Td-pur® and Boostrix® dTpa vaccines used in this study are commercially available in Switzerland and will be purchased for the study. One batch of each vaccine will be used for the entire study.

All vaccines are presented in 0.5 mL pre-filled syringes to be administered by intramuscular injection. The study vaccine Pertagen® and Boostrix® dTpa will be administered in the non-dominant deltoid. If applicable, Td-pur® will be administered in the contralateral deltoid.

At Day 0, eligible subjects will be randomized in a 1:1 ratio into one of the following vaccine groups:

Group 1 Pertagen® and Td-pur 30 volunteers Group 2 Boostrix® dTpa 30 volunteers

A randomization list containing subject numbers and vaccine group assignments will be established and provided to the clinical investigators. Each participant will be immunized according to the vaccine group assignment. At study site, the Principal investigator will designate the blinded and unblinded teams in order to keep the observer-blind design of the study.

The unblinded personal will be responsible for study vaccine preparation, handling, storage and accountability, and immunization.

The blinded team will be responsible for assessing adverse events. The laboratory staff performing the immunological assays will also be blinded. After vaccination, volunteers will be observed for 30 minutes at study site for any immediate post-immunization reactions. Reactogenicity and safety will be assessed during study visits at the clinical trial unit (CTU) on Day 0 and Day 28 after immunization. At Day 0 (Visit 1, vaccination day), a Diary Card will be distributed to study volunteer to record post-immunization local and systemic reactions and adverse events. At Day 28 (Visit 2), investigator will reconcile and transcribe the Diary Card information in the CRF. Post-immunization local and systemic reactions will be collected and monitored for 7 days after vaccination. All adverse events, including SAEs, will be collected and monitored for 28 days after vaccination (until Visit 2).

Study participants will be contacted by phone at Day 7 to confirm that adverse reactions have subsided. Should this not be the case, an unscheduled visit will be considered as appropriate.

All AEs and SAEs occurring within the 28 days following treatment and observed by the Investigator or reported by the volunteer, whether or not attributed to study intervention, will be recorded in the CRF. All AEs that result in a volunteer's withdrawal from the study will be followed up until a satisfactory resolution occurs, or until a non-study related causality is assigned (if the volunteer consents to this).

Sample size calculation This is a phase II randomized, observer-blind controlled pilot study to compare the safety and immunogenicity of acellular pertussis vaccines including chemically or genetically-detoxified pertussis toxin in adolescents previously immunized with acellular vaccines. The sample size for this study is based on clinical and practical considerations and not on a formal statistical power calculation. Where applicable, 2-sided test at the 5% significance level will be utilized with no multiplicity adjustment. P-values will be considered exploratory only. Sixty volunteers will be randomized in total, with 30 in each group.

Safety analysis The safety analysis will include all randomized subjects who have received a dose of study vaccine.

The overall percentage of subjects with at least one spontaneously reported adverse event, with date of onset up to 28 days after vaccination will be tabulated with exact 95% confidence intervals, by type of adverse event; by severity; and by causality. They will be displayed by vaccine group as both frequencies and percentages on the ITT data set.

All reported adverse events that start post-vaccination will be tabulated. If a given disease is already reported as ongoing at the first visit on the medical history pages, it will be counted and tabulated as a vaccine emergent adverse event only if it worsens after the immunization with the study vaccine.

Serious adverse events and discontinuation due to adverse event(s) will be described in detail by vaccine group.

Immunogenicity analyses The primary immunogenicity endpoint will assess the immune response to Pertagen® - as compared to Boostrix® dTpa - by measuring the Day 28 geometric mean concentration (GMC) of neutralizing antibodies to PT.

The other immunogenicity end-points include:

* GMCs of PT, FHA, tetanus and diphtheria-toxoid specific IgG antibodies measured by ELISA
* Seroresponse rates of PT, FHA, tetanus and diphtheria-toxoid specific IgG antibodies measured by ELISA
* Reverse cumulative distribution curves of PT neutralizing antibodies, and of PT, FHA, tetanus and diphtheria-toxoid IgG antibodies
* To compare PT-specific responses elicited by Pertagen® in adolescents previously immunized (this study) or not (BioNet Phase II/III TDA202) by acellular pertussis vaccines The following descriptive statistics will be provided for each variable: number of subjects, percentages, mean, geometric mean, standard deviation, median, minimum, maximum, and range.

Quality Control and Quality Assurance Procedure Approved site-specific SOPs will be used at clinical and laboratory sites. Monitoring will be performed according to ICH Good Clinical Practice (GCP) by the Centre de Recherche Clinique (CRC) of the University Hospital of Geneva. Following a Monitoring Plan and written SOPs, the monitors will verify that the clinical trial is conducted and data are generated, documented and reported in compliance with the protocol, GCP and the applicable regulatory requirements. The CTU will provide direct access to all trial-related source data, documents and reports for the purpose of monitoring and inspection by local and regulatory authorities.

ELIGIBILITY:
Inclusion criteria

The volunteer must satisfy the following criteria to be eligible for the study:

1. Has provided written informed consent before enrollment;
2. Male or female, ages 11-15 years (inclusive) at the time of enrollment;
3. With documented history of acellular pertussis immunization (5 doses);
4. Free of clinically significant health problems, as determined by pertinent medical history and clinical examination at study screening;
5. Non-pregnant, non-lactating female :

   * for female subjects who had menarche, this implies a negative urinary pregnancy test at enrolment;
   * If sexually active, female subjects must be willing to use reliable birth control measures for 1 month after vaccination;
6. Able to attend all scheduled visits and to understand and comply with the study procedures; Exclusion criteria

The volunteer may not enter the study if any of the following apply:

1. Prior dTpa immunization within the last 5 years or prior dT immunization within the last 2 years, or any other investigational vaccine likely to impact on interpretation of the trial data, as judged by the Principal Investigator;
2. Suspected or confirmed pertussis infection within the last 10 years or documented pertussis infection in a household member within the last 10 years;
3. History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions;
4. Known hypersensitivity or allergy to diphtheria, tetanus, or pertussis vaccine (including excipients);
5. Receipt of investigational product up to 30 days prior to enrollment or ongoing participation in another interventional clinical trial;
6. Receipt of licensed vaccines within 30 days of planned study immunization or ongoing participation in another clinical interventional trial;
7. Acute or chronic, clinically significant psychiatric, hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the Investigator based on medical history, physical exam;
8. Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection, asplenia, cytotoxic therapy in the previous 5 years, and/or diabetes;
9. Any chronic or active neurologic disorder, including seizures, and epilepsy, excluding febrile seizures as a child;
10. Has a known history of Guillain-Barré Syndrome;
11. Has an active malignancy or recent (<10 years) history of metastatic or hematologic malignancy;
12. Suspected or known alcohol and/or illicit drug abuse within the past 5 years;
13. Pregnant or lactating female, or female who intends to become pregnant during the study period;
14. Administration of immunoglobulins and/or any blood products within the 120 days preceding study entry or planned administration during the study period;
15. Receipt of chronic (>14 days) immunosuppressants or other immune modifying drugs within 6 months of study entry:

    * For corticosteroids, this will mean prednisone or equivalent ≥0.5 mg/kg/day,
    * Intranasal and topical steroids are allowed;
16. Any other significant finding that, in the opinion of the investigator, would increase the risk of the individual's having an adverse outcome by participating in this study.

Temporary exclusion criteria at the time of randomization

The following criteria constitute contraindications to administration of vaccine at that point in time; if any one of these occurs at the time scheduled for randomization, the subject may be randomized at a later date without the need for re-screening, at the discretion of the Investigator, or withdrawn at the discretion of the Investigator:

* Acute disease at the time of randomization. (Acute disease in the context of this trial is defined as the presence of a moderate or severe illness with or without fever.) The vaccine/placebo can be administered to persons with a minor illness such as mild upper respiratory tract infection with or without low-grade febrile illness, i.e. temperature of ≤37.5°C;
* Body temperature ≥38°C within 3 days of the intended vaccination;
* Any other significant finding that, in the opinion of the investigator, would temporarily increase the risk of the individual's having an adverse outcome by participating in this study.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-10-27 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
Geometric mean concentration (GMC) of neutralizing antibodies to PT | At 28 days after vaccination

SECONDARY OUTCOMES:
Safety endpoints evaluated by solicited local and systemic reactions and unsolicited adverse events (AEs) | Solicited local and systemic reactions will be followed up for 7 days and AEs for 28 days after vaccination
GMCs and seroresponse rates of PT, FHA, tetanus and diphtheria-toxoid specific IgG antibodies measured by ELISA | At 28 days after vaccination
Seroresponse rates of PT specific neutralizing antibodies Time Frame: At 28 days after vaccination | At 28 days after vaccination
Reverse cumulative distribution curves of PT neutralizing antibodies, and of PT, FHA, tetanus and diphtheria-toxoid IgG antibodies | At 28 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Claire-Anne Siegrist, MD, Principal Investigator — Center for Vaccinology, Medical Faculty (UNIGE) and University Hospitals of Geneva (HUG), CMU
Locations (1):
- Pediatric clinical trial platform, University Hospitals of Geneva City: Geneva, Geneva, Switzerland

REFERENCES:
- [Background] Buasri W, Impoolsup A, Boonchird C, Luengchaichawange A, Prompiboon P, Petre J, Panbangred W. Construction of Bordetella pertussis strains with enhanced production of genetically-inactivated Pertussis Toxin and Pertactin by unmarked allelic exchange. BMC Microbiol. 2012 Apr 23;12:61. doi: 10.1186/1471-2180-12-61. PMID 22524455
- [Background] Ibsen PH. The effect of formaldehyde, hydrogen peroxide and genetic detoxification of pertussis toxin on epitope recognition by murine monoclonal antibodies. Vaccine. 1996 Apr;14(5):359-68. doi: 10.1016/0264-410x(95)00230-x. PMID 8735545
- [Background] Podda A, Carapella De Luca E, Titone L, Casadei AM, Cascio A, Bartalini M, Volpini G, Peppoloni S, Marsili I, Nencioni L, et al. Immunogenicity of an acellular pertussis vaccine composed of genetically inactivated pertussis toxin combined with filamentous hemagglutinin and pertactin in infants and children. J Pediatr. 1993 Jul;123(1):81-4. doi: 10.1016/s0022-3476(05)81543-4. PMID 8320630
- [Background] Rappuoli R. The vaccine containing recombinant pertussis toxin induces early and long-lasting protection. Biologicals. 1999 Jun;27(2):99-102. doi: 10.1006/biol.1999.0189. PMID 10600193
- [Background] Salmaso S, Mastrantonio P, Tozzi AE, Stefanelli P, Anemona A, Ciofi degli Atti ML, Giammanco A; Stage III Working Group. Sustained efficacy during the first 6 years of life of 3-component acellular pertussis vaccines administered in infancy: the Italian experience. Pediatrics. 2001 Nov;108(5):E81. doi: 10.1542/peds.108.5.e81. PMID 11694665
- [Derived] Blanchard Rohner G, Chatzis O, Chinwangso P, Rohr M, Grillet S, Salomon C, Lemaitre B, Boonrak P, Lawpoolsri S, Clutterbuck E, Poredi IK, Wijagkanalan W, Spiegel J, Pham HT, Viviani S, Siegrist CA. Boosting Teenagers With Acellular Pertussis Vaccines Containing Recombinant or Chemically Inactivated Pertussis Toxin: A Randomized Clinical Trial. Clin Infect Dis. 2019 Mar 19;68(7):1213-1222. doi: 10.1093/cid/ciy594. PMID 30759183